CLINICAL TRIAL: NCT03186326
Title: Multicenter Randomized Phase II Study Comparing the Effectiveness and Tolerance of Avelumab Versus Standard 2nd Line Treatment Chemotherapy in Patients With Colorectal Metastatic Cancer With Microsatellite Instability (MSI)
Brief Title: Standard Chemotherapy vs Immunotherapie in 2nd Line Treatment of MSI Colorectal Mestastatic Cancer
Acronym: SAMCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 54 - FFCD 1603
Record Dates: First submitted 2017-05-17; First posted 2017-06-14 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Colorectal Cancer; MSI
Keywords: immunotherapy; second line
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; IFL protocol; avelumab; Panitumumab; Cetuximab; Bevacizumab; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Chemotherapy (standard treatment) (Active Comparator): FOLFOX or FOLFIRI +/- targeted therapy
  Interventions: Drug: FOLFOX regimen; Drug: FOLFIRI Protocol; Drug: Panitumumab; Drug: Cetuximab; Drug: Bevacizumab; Drug: Aflibercept
- Arm B - Immunotherapy (experimental arm) (Experimental): Avelumab
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: FOLFOX regimen — A course of treatment every 14 days
  Oxaliplatin: 85 mg/m² IV over 2 hours Folinic acid: 400 mg/m² (or 200 mg/m² if Elvorine) IV over 2 hours 5FU bolus: 400 mg/m² IV bolus over 10 minutes in 100 ml 0.9% NaCl 5FU continuous: 2,400 mg/m² in NaCl 0.9% in IV over 46 hours
  Arms: Arm A Chemotherapy (standard treatment)
Drug: FOLFIRI Protocol — A course of treatment every 14 days
  Irinotecan: 180 mg/m² IV over 1H30 Folinic acid: 400 mg/m² (or 200 mg/m² if Elvorine) IV over 2 hours 5FU bolus: 400 mg/m² IV bolus over 10 minutes in 100 ml 0.9% NaCl 5FU continuous: 2,400 mg/m² in NaCl 0.9% in IV over 46 hours
  Arms: Arm A Chemotherapy (standard treatment)
Drug: Avelumab — A course of treatment every 14 days. Premedication obligatory with antihistamines and paracetamol (example: 25-50 mg diphenhydramine and 500-650 mg paracetamol) IV, approximately 30 to 60 minutes before each dose of avelumab.
  Then:
  Avelumab: 10 mg/kg IV in 1 hour diluted with 0.9% saline solution; alternatively a 0.45% saline solution can be used if needed
  Arms: Arm B - Immunotherapy (experimental arm)
Drug: Panitumumab — Administered at 6 mg/Kg
  Arms: Arm A Chemotherapy (standard treatment)
Drug: Cetuximab — Administered at 500 mg/m²
  Arms: Arm A Chemotherapy (standard treatment)
Drug: Bevacizumab — Administered at 5 mg/Kg
  Arms: Arm A Chemotherapy (standard treatment)
Drug: Aflibercept — Administered at 4 mg/Kg
  Arms: Arm A Chemotherapy (standard treatment)

SUMMARY:
Immune chekpoints (ICI) are evaluated in many digestive cancers. Certain types of cancer appear to be rather refractory to ICI such as colorectal cancers (CRC). However, the MSI CRC representing approximately 15% of the CRCs exhibits a high mutational load which generates many potentially immunogenic neoantigens. In addition, strong expression of PD-L1 was found in the MSI CRCs relative to the CRC (MSS) stages. Localized MSI CRCs have a better prognosis than MSS CRCs, probably due to immunogenic neoantigens associated with a CD8 + T-specific immune response. On the oher hand, in metastatic CRC (mCRC) things are different because i) the MSI frequency is only 4 to 7% and ii) the good prognosis conferred by the MSI status is controversial.

Preliminary results suggest that patients with MSI mCRC are highly sensitive to ICI even chemoresistant tumors receiving several lines of chemotherapy. Recently, another anti-PD1 alone or in combination with an anti-CTLA4 (antigen associated with cytotoxic T-lymphocyte 4) was tested in the MSI CRCs and a selection of interesting results in heavily pretreated patients with a disease control rate of 56% for monotherapy and 81% for combinated therapy.

Anti-PD1s now have marketing authorization for patients with melanoma and metastatic pulmonary carcinoma , Which are known to have a high level of mutations . ICIs appear to be as promising in MSI CRCs as in other tumors and therefore face the same major challenges.

Avalumab is an anti-PD-L1 antibody recently tested in several different types of tumors with promising results and is currently being studied in phase III in gastric cancer. There is no data on the effectiveness of this ICI in the MSI mCRCs. In addition, only anti-PD1 was used in the MSI-mCRC and not the anti-PD-L1, and only in chemoresistance (3rd line or more). The main objective of the SAMCO study is to test the efficacy and tolerance of avelumab in the 2nd line of treatment in patients with a MSI mCRC progression after standard 1st line chemotherapy +/- targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma with metastasis(es) non-resectable
* MSI-H determined by immunohistochemistry (loss of expression of MLH1, MSH2, MSH6 and/or PMS2) or by molecular biology
* At least one measurable target (primary tumor or metastasis) according to RECIST v1.1
* Mutational status RAS and BRAF
* Age ≥ 18
* OMS ≤ 2
* Life expectancy < 3 months
* Patient failure (progression or unacceptable toxicity) of chemotherapy containing fluoropyrimidine (capecitabine or 5FU) +/- irinotecan +/- oxaliplatin with or without cetuximab, bevacizumab and panitumumab (patients in progression during or within 3 months after discontinuation of adjuvant chemotherapy are eligible)
* PNN > 1500/mm3, platelets > 100 000/mm3, Hb > 9 g/dL
* Total bilirubin < 25 µmol/L, ASAT < 5x LSN, ALAT < 5 x LSN, PT > 60%, , PAL<2.5 x LSN ( < 5 x LSN in case of hepatic metastasis)
* Creatinine clearance > 50 ml/min according to MDRD formula (≥ 30 ml/min according to the Cockcroft-Gault formula)
* Patient belonging to a social security scheme
* Patient information and signature of the informed consent

Exclusion Criteria:

* Patient immediately eligible for a curative therapy (surgical and/or percutaneous) after discussion in CPR
* Patient treated with FOLFIRINOX or FOLFOXIRI in 1st line
* Cerebral metastasis
* Previous treatment with anti-PD1 or anti-PDL1
* Autoimmune disease that might be aggravated during treatment with an immuno-stimulating agent (patients with type I diabetes, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible)
* Immunosuppressive long-term treatment (patients necessitating a corticotherapy are eligible if they are administered in doses < or = to the equivalent of 10 mg of prednisone daily, administration of steroids by a route resulting in minimal systemic exposure (local, intra-anal, intraocular or inhalation) are eligible).
* Transplant patients (including stem cell transplants), HIV positive or other immune deficiency syndromes
* Active infection by HBV or HCV
* Known severe hypersensitivity to monoclonal antibodies or history of anaphylactic shock, or uncontrolled asthma
* Any known specific contraindication or allergy to the treatments used in the study
* Persistence of toxicities related to 1st line chemotherapy grade > 2 (NCI-CTC v4.0) (except alopecia and neuropathy sequelae of oxaliplatin)
* Vaccination during the 4 weeks preceding the start of treatment
* Known deficit in DPD
* QT/QTc interval > 450 msec for men and > 470 msec for women
* K+ < LIN, Mg2+ < LIN, Ca2+ < LIN
* Following alterations in the 6 months prior to inclusion: myocardial infarction, angina, severe/unstable angina, coronary artery bypass surgery, congestive heart failure NYHA class II, III or IV, stroke or transient ischemic attack
* Any progressive pathology not stabilised over the past 6 months: hepatic failure, renal failure, respiratory failure
* Patient with interstitial pneumonitis or pulmonary fibrosis
* History of chronic diarrhea or inflammatory disease of the colon or rectum, or unresolved occlusion or sub-occlusion in symptomatic treatment
* History of malignant pathologies during the past 5 years except basocellular skin carcinoma or in situ cervical carcinoma, properly treated
* Patient already included in another clinical trial during treatment with an experimental molecule for L2
* Lack of effective contraception in patients (men and/or women) of childbearing age, pregnant or breastfeeding women, women of childbearing age not having had a pregnancy test
* Persons deprived of liberty or under supervision
* Impossibility of undergoing medical monitoring during the trial for geographic, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) according to the investigator | up to 12 months
  Progression is defined as RECIST v1.1 criteria. Death is also considered as an event

SECONDARY OUTCOMES:
Overall Survival | up to 60 months
  Defined as death due to all causes

CONTACTS AND LOCATIONS:
Overall Officials: Julien Taieb, Pr, Principal Investigator — HOPITAL EUROPEEN G. POMPIDOU
Locations (120):
- France (120):
  - Ch - Centre Hospitalier D'Abbeville, Abbeville
  - Ch - Centre Hospitalier Du Pays D'Aix, Aix-en-Provence
  - Chu - Hôpital Sud - Service D'Hge, Amiens
  - Privé - Clinique de L'Europe, Amiens
  - Cac - Ico Site Paul Papin, Angers
  - CHU - Hôtel Dieu, Angers
  - Privé - Hopital Privé D'Antony, Antony
  - Ch - Hôpital Victor Dupouy, Argenteuil
  - Ch - Centre Hospitalier Ardeche Meridionale, Aubenas
  - Ch - Ght Unyon Auxerre, Auxerre
  - Ch - Hôpital Henri Duffaut, Avignon
  - Privé - Institut Sainte Catherine, Avignon
  - Ch - Centre Hôspitalier Côte Basque, Bayonne
  - Ch - Centre Hospitalier de Beauvais, Beauvais
  - Chu - Jean Minjoz, Besançon
  - Privé - Centre de Radiotherapie Pierre Curie, Beuvry
  - Privé - Polyclinique Bordeaux Nord, Bordeaux
  - Privé - Cac Institut Bergionié, Bordeaux
  - Privé - Polyclinique Saint-Privat, Boujan-sur-Libron
  - Ch - Hôpital Duchenne, Boulogne-sur-Mer
  - Privé - Clinique Pasteur Lanroze Cfro, Brest
  - Privé - Centre Maurice Tubiana, Caen
  - Privé - Cac Centre Francois Baclesse, Caen
  - Privé - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Ch - Centre Hospitalier de Carcassonne, Carcassonne
  - Chi - Centre Hospitalier de Castres Mazamet, Castres
  - Ch - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Privé - Hopital Prive Sainte Marie, Chalon-sur-Saône
  - Ch - Centre Hospitalier Metropole Savoie, Chambéry
  - Ch - Centre Hospitalier de Charleville Mezieres, Charleville
  - Ch - Centre Hospitalier General, Châlons-en-Champagne
  - Ch - Centre Hospitalier de Châteauroux, Châteauroux
  - Ch - Centre Hospitalier de Cholet, Cholet
  - Ch - Hopitaux Civils de Colmar, Colmar
  - Privé - Clinique Saint Come, Compiègne
  - Ch - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Privé - Clinique Des Cèdres, Cornebarrieu
  - Privé - Clinique de Flandre, Coudekerque-Branche
  - Ch - Ghpso Site de Creil, Creil
  - Ch - Chic de Créteil, Créteil
  - Chu - Aphp - Hopital Henri Mondor, Créteil
  - Privé - Institut de Cancerologie de Bourgogne Grrecc, Dijon
  - Chu - Hopital Francois Mitterrand, Dijon
  - Privé - Cac- Centre Georges-Francois Leclerc, Dijon
  - Privé - Ghm Institut Daniel Hollard, Grenoble
  - Chu - Grenoble Alpes, Grenoble
  - Privé - Clinique Sainte Marguerite, Hyères
  - Ch - Centre Hospitalier Marne La Vallee-Jossigny, Jossigny
  - Chd - Centre Hospitalier Vendee, La Roche-sur-Yon
  - Privé - Clinique Du Cap D'Or, La Seyne-sur-Mer
  - Ch - Hopital Andre Mignot, Le Chesnay
  - Ch - Hopital Louis Pasteur - Oncologie Hematologie, Le Coudray
  - Privé - Cmc Les Ormeaux, Le Havre
  - Chu - Aphp - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Ch - Centre Hospitalier Du Mans, Le Mans
  - Ch - Centre Hospitalier Docteur Schaffner, Lens
  - Ch - Hôpital Franco Britannique, Levallois-Perret
  - Privé - Cac - Centre Oscar Lambret, Lille
  - Chu - Dupuytren, Limoges
  - Ch - Gh Nord Essone, Longjumeau
  - Chu - Hôpital de La Croix Rousse, Lyon
  - Privé - Cac Centre Léon Berard, Lyon
  - Chu - Hôpital Edouard Herriot, Lyon
  - Privé - Cac Institut Paoli Calmettes, Marseille
  - Ch - Hôpital Saint Joseph, Marseille
  - Privé - Hôpital Européen Marseille, Marseille
  - Chu - La Timone, Marseille
  - Ch - Ghi de L'Est Francilien Site de Meaux, Meaux
  - Ch - Hôpital Belle Isle, Metz
  - Privé - Clinique Claude Bernard, Metz
  - Ch - Hôpital Layné, Mont-de-Marsan
  - Ch - Centre Hospitalier de Montceau Les Mines, Montceau-les-Mines
  - Ch - Centre Hospitalier de Montélimar, Montélimar
  - Ch - Groupe Hospitalier Intercommunal Le Raincy, Montfermeil
  - Privé - Centre de Cancérologie Du Grand Montpellier, Montpellier
  - Privé - Hôpital Prive Du Confluent Sas, Nantes
  - Privé - Cac - Centre Antoine Lacassagne, Nice
  - Chu - Hôpital Caremeau, Nîmes
  - Chr - Centre Hospitalier Régional de La Source, Orléans
  - Privé - Cac - Institut Curie, Paris
  - Chu - Hôpital Cochin, Paris
  - Chu - Hôpital Europeen Georges Pompidou, Paris
  - Chu - Aphp - Hôpital Saint Louis, Paris
  - Chu - Hôpital Saint Antoine, Paris
  - Chu - Aphp - Gh La Pitié Salpêtrière, Paris
  - Ch - Centre Hospitalier de Pau, Pau
  - Ch - Hôpital Saint Jean, Perpignan
  - Chu - Hôpital Haut Lévêque, Pessac
  - Privé - Polyclinique Francheville, Périgueux
  - Ch - Hôpital Lyon Sud, Pierre-Bénite
  - Privé - Centre Cario - Hcpa, Plérin
  - Chu - Hôpital de La Miletrie, Poitiers
  - Ch - Hôpital Rene Dubos, Pontoise
  - Ch - Hôpital Annecy Genevois, Pringy
  - Ch - Chic - Centre Hospitalier de Cornouaille, Quimper
  - Chu - Hôpital Robert Debre, Reims
  - Chu - Centre Hospitalier Universitaire Pontchaillou, Rennes
  - Privé - Centre de Radiotherapie Et D'Oncologie Médicale de L'Essone, Ris-Orangis
  - Privé - Clinique Pasteur, Ris-Orangis
  - Ch - Hôpitaux Drome Nord, Romans-sur-Isère
  - Chu - Hôpital Charles Nicolle, Rouen
  - Privé - Hôpital Privé Saint Gregoire, Saint-Grégoire
  - Privé - Clinique de L'Union, Saint-Jean
  - Privé - Cmco Côte D'Opale, Saint-Martin-Boulogne
  - Privé - Clinique Mutualiste de L'Estuaire - Cite Sanitaire, Saint-Nazaire
  - Chu - Hôpital Nord - Saint-Étienne, Saint-Priest-en-Jarez
  - Privé - Clinique Trenel, Sainte-Colombe
  - Ch - Centre Hospitalier de Soisson, Soissons
  - Ch - Centre Hospitalier de Saint-Malo, St-Malo
  - Privé - Cac - Institut de Cancérologie de Strasbourg Europe, Strasbourg
  - Privé - Clinique Sainte Anne, Strasbourg
  - Ch - Hopitaux Du Leman, Thonon-les-Bains
  - Ch - Hôpital Sainte Musse, Toulon
  - Chu - Hôpital Rangueil, Toulouse
  - Chu - Hôpital Trousseau, Tours
  - Chu - Hôpital Nancy-Brabois, Vandœuvre-lès-Nancy
  - Privé - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Chu - Aphp - Hôpital Paul Brousse, Villejuif
  - Privé - Cac - Gustave Roussy, Villejuif
  - Ch - Centre Hospitalier Intercommunal, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Taieb J, Andre T, El Hajbi F, Barbier E, Toullec C, Kim S, Bouche O, Di Fiore F, Chauvenet M, Perrier H, Evesque L, Laurent-Puig P, Emile JF, Bez J, Lepage C, Tougeron D. Avelumab versus standard second line treatment chemotherapy in metastatic colorectal cancer patients with microsatellite instability: The SAMCO-PRODIGE 54 randomised phase II trial. Dig Liver Dis. 2021 Mar;53(3):318-323. doi: 10.1016/j.dld.2020.11.031. Epub 2020 Dec 25. PMID 33359404
- [Derived] Taieb J, Sullo FG, Lecanu A, Bourreau C, Barbier E, Gandini A, Bez J, Mulot C, Di Fiore F, Elhajbi F, Borg C, Bouche O, Aparicio T, Zaanan A, Andre T, Tougeron D, Taly V, Laurent-Puig P. Early ctDNA and Survival in Metastatic Colorectal Cancer Treated With Immune Checkpoint Inhibitors: A Secondary Analysis of the SAMCO-PRODIGE 54 Randomized Clinical Trial. JAMA Oncol. 2025 Aug 1;11(8):874-882. doi: 10.1001/jamaoncol.2025.1646. PMID 40531517
- [Derived] Taieb J, Bouche O, Andre T, Le Malicot K, Laurent-Puig P, Bez J, Toullec C, Borg C, Randrian V, Evesque L, Corbinais S, Perrier H, Buecher B, Di Fiore F, Gallois C, Emile JF, Lepage C, Elhajbi F, Tougeron D; SAMCO-PRODIGE 54 Investigators. Avelumab vs Standard Second-Line Chemotherapy in Patients With Metastatic Colorectal Cancer and Microsatellite Instability: A Randomized Clinical Trial. JAMA Oncol. 2023 Oct 1;9(10):1356-1363. doi: 10.1001/jamaoncol.2023.2761. PMID 37535388